CLINICAL TRIAL: NCT07003243
Title: Effectiveness of Topical Application of Melatonin On Bone Density and Implant Stability In Immediate Implantation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali Mohammed Ali, Doctor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Melatonin in immediate implant
Record Dates: First submitted 2025-05-20; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Immediate Implant Placement; Melatonin Production

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Participants receive bone graft + saline only
- Study group (Experimental): Participants receive bone graft + 3 mg melatonin + saline
  Interventions: Drug: Local melatonin powder

INTERVENTIONS:
Drug: Local melatonin powder — A single topical dose of 3 mg of pure melatonin powder was mixed with particulate bone graft and normal saline, then packed into the jumping gap around immediately placed dental implants. The intervention was performed at the time of surgery following atraumatic tooth extraction. The aim was to enhance osseointegration and minimize crestal bone loss over a 6-month healing period.
  Arms: Study group

SUMMARY:
Dental implants have revolutionized the replacement of missing teeth, offering predictable and long-lasting rehabilitation for both fully and partially edentulous patients. Since Brånemark's landmark work in 1969, which defined osseointegration as "a direct structural and functional connection between ordered living bone and the surface of a load-bearing implant" (Brånemark et al., 1969), implantology has become an integral part of restorative dentistry.

Traditionally, implant therapy followed a delayed protocol requiring a healing period of up to six months after extraction to allow complete soft and hard tissue regeneration before implant placement (Adell et al., 1981). This approach was based on the belief that mature bone is essential for achieving osseointegration. However, subsequent research demonstrated that immediate placement of implants into fresh extraction sockets can also lead to successful osseointegration without compromising outcomes (Araujo et al., 2005).

Immediate implant placement, defined as placing an implant at the time of tooth extraction, has gained popularity due to its clinical benefits. These include a reduction in surgical sessions, shortened overall treatment time, preservation of the alveolar ridge, especially the buccal plate, and superior soft tissue esthetics (Van Der Weijden et al., 2009). However, these advantages are contingent upon achieving primary implant stability and proper case selection. A biological challenge that often arises in such cases is the presence of a "jumping gap" - a void between the implant surface and the socket wall - which may require the use of bone grafts or regenerative materials to facilitate bone fill and stability.

In recent years, research has explored various biologically active molecules and growth factors to enhance bone healing and implant integration, especially in immediate placement protocols. These include bone morphogenetic proteins (BMPs), platelet-rich plasma (PRP), and platelet-derived growth factors. Among these, melatonin has emerged as a promising agent due to its multifaceted biological activity (Zechner et al., 2003).

Melatonin (N-acetyl-5-methoxytryptamine) is an endogenously produced neurohormone primarily secreted by the pineal gland. While best known for regulating circadian rhythms, melatonin also possesses strong antioxidant, anti-inflammatory, and bone-promoting properties. It enhances osteoblast proliferation, stimulates collagen matrix formation, and inhibits osteoclast-mediated bone resorption. These effects make melatonin a potential therapeutic agent for improving bone density and implant stability.

Topical application of melatonin at implant sites has shown encouraging results in experimental models, demonstrating improved bone-to-implant contact, accelerated bone regeneration, and enhanced mechanical stability. These findings suggest a potential role for melatonin in immediate implant protocols, where rapid healing and early osseointegration are critical for clinical success.

Given the biological potential of melatonin, the present study aims to evaluate the effectiveness of topical application of melatonin on bone density and implant stability in immediate implantation cases through a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Presence of single-rooted non-restorable anterior or premolar teeth indicated for extraction.
* Jumping gap ≥ 2 mm as measured clinically or radiographically.
* Apical bone ≥ 2 mm beyond the socket on radiographs.
* Good general health with no contraindications for oral surgery.
* Patient willing to undergo immediate implant placement.
* Ability and willingness to return for follow-up visits.
* Provided written informed consent.

Exclusion Criteria:

* Presence of active periodontal disease or acute infection at the surgical site.
* Patients with systemic conditions that could compromise healing (e.g., uncontrolled diabetes, immune compromise).
* History of bisphosphonate therapy.
* Head and neck irradiation.
* Pregnancy or lactation.
* Heavy smokers (≥20 cigarettes/day).
* -Bruxism or parafunctional habits.
* Inability to comply with study protocol or follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in crestal bone level around dental implants | Baseline (Day 0) and 6 months postoperatively
  Radiographic measurement of vertical crestal bone loss using cone-beam computed tomography (CBCT) at baseline and after 6 months to assess the effect of topical melatonin application on bone preservation.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No